CLINICAL TRIAL: NCT05241028
Title: Adjuvant Therapy of Ensatinib in Patients With Stage IB-IIIA ALK-positive Non-small Cell Lung Cancer: a Prospective, Multi-center, Single-arm Exploratory Study
Brief Title: Adjuvant Therapy of Ensartinib in Stage IB-IIIA ALK-positive Non-small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hebei Medical University Fourth Hospital (Other)
Responsible Party: Principal Investigator, LiuJunFeng, Director of thoracic surgery, Hebei Medical University Fourth Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BD-EN-IV006
Record Dates: First submitted 2022-01-24; First posted 2022-02-15 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Ensartinib; adjuvant therapy; ALK; Tyrosine kinase inhibitor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — ensartinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ensartinib (Experimental): Ensartinib 225mg oral daily for 3 years or until recurrence of the disease or intolerable toxicity
  Interventions: Drug: Ensartinib

INTERVENTIONS:
Drug: Ensartinib — Ensartinib 225mg oral daily for 3 years or until recurrence of the disease or intolerable toxicity
  Other Names: X-396 capsule

SUMMARY:
This is a prospective, multi-center, single-arm, phase 2 study aiming to assess the efficacy and safety of adjuvant use of Ensartinib in stage IB-IIIA non-small cell lung cancer (NSCLC) with positive ALK-fusion. Enrolled patients will take Ensatinib for 3 years or until recurrence of the disease or intolerable toxicity, following complete tumour resection with or without adjuvant standard chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Completely resected pathological stage IB-IIIA NSCLC with ALK-fusion positive (confirmed by FISH, IHC or NGS).
* Males or females aged ≥18 years, ≤75 years.
* ECOG performance status 0-2.
* Completely recovered from surgery or standard postoperative chemotherapy before receiving adjuvant ensatinib treatment. (When starting the study treatment, the patient must have recovered from all toxicities greater than CTCAE Grade 1 caused by the previous treatment, except for hair loss and Grade 2 neuropathy related to previous platinum-based treatments).
* Clinical examinations before treatment report no signs of disease recurrance.
* With enough tumor histology specimens (non-cytology) for molecular marker analysis.
* hemoglobin concentration ≥ 100 g/L (permit to maintain hematologic criteria by blood transfusion); absolute neutrophil count (ANC) ≥1.5×10^9/L; platelet count ≥100×10^9/L.
* Liver Function: TBil ≤2xULN; ALT and AST ≤2.5xULN;
* Renal Function: Cr ≤1.5xULN, and Ccr ≥60ml/min;
* Signed inform consent form by patient or his/her legal representative.
* Comply with study protocol and procedure, and be able to take oral medication.
* Female patients of childbearing potential must have a negative urine pregnancy test within 7 days before study treatment.
* Eligible patients of reproductive potential (both sexes) must agree to use a reliable method of birth control before enrollment, during the study period and for at least 8 weeks after their last dose of study therapy.

Exclusion Criteria:

* Having targeted medication therapy (including tyrosine kinase inhibitor or monoclonal antibody) and experimental therapy for NSCLC in the past.
* Having local radiotherapy of NSCLC.
* Known allergy to Ensatinib or any of the ingredients in this product.
* Previously suffering from interstitial lung disease, drug-induced interstitial disease, radiation pneumonia that requires hormone therapy, or any clinically evidenced active interstitial lung disease; CT scan at baseline revealed the presence of idiopathic pulmonary fibrosis.
* Any unstable systemic disease, including: active infection, uncontrolled high blood pressure, unstable angina pectoris, angina pectoris that started within the last 3 months, congestive heart failure (≥ New York Heart Association [NYHA] II Grade), myocardial infarction (6 months before enrollment), severe arrhythmia requiring medical treatment; liver, kidney or metabolic diseases.
* Women who are pregnant or breastfeeding.
* Having history of neurological or psychiatric disorders, including epilepsy or dementia.
* Other conditions investigators evaluate that patient is not eligible to this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
3-year disease free survival rate (DFSR) | 3 years
  Defined as the percentage of patients alive and disease free at 3 years

SECONDARY OUTCOMES:
5-year overall survival rate | 5 years
  Defined as the percentage of patients alive at 5 years
disease free survival (DFS) | Up to 5 years
  Defined as the time from the date of starting treatment until the date of disease recurrence or death (by any cause in the absence of recurrence)
overall survival (OS) | Up to 5 years
  Defined as the time from starting treatment to death.
Adverse Events | Up to 3 years
  The safety and tolerability profile of Ensartinib

CONTACTS AND LOCATIONS:
Locations (1):
- Jun Feng Liu, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: No